CLINICAL TRIAL: NCT07395128
Title: Lateral Plantar Artery Embolization to Treat Pain Chronic Heel Pain Due To Plantar Fasciitis A Pilot Study to Assess Feasibility
Brief Title: Lateral Plantar Artery Embolization For Plantar Fasciitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joint & Vascular Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1402856
Record Dates: First submitted 2026-01-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Plantar Fasciitis, Chronic; Plantar Fasciitis
Keywords: plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Lateral Plantar Artery Embolization (Experimental)
  Interventions: Device: Lipiodol

INTERVENTIONS:
Device: Lipiodol — Participants will receive a transcatheter arterial embolization of the lateral plantar artery branches. The intervention involves the selective catheterization of the calcaneal branches under fluoroscopic guidance using a microcatheter. A mixture of Lipiodol (a transient liquid embolic agent) and iodinated contrast media is injected until an endpoint of "near stasis" is reached. A maximum of 5 mL of Lipiodol will be used per procedure. This intervention specifically targets the hypervascularity (neovascularization) associated with chronic plantar fasciitis to alleviate pain and reduce inflammation.

SUMMARY:
The goal of this clinical trial is to learn if lateral plantar artery embolization using Lipiodol can safely and effectively treat chronic heel pain due to plantar fasciitis in adults aged 25 to 80. The main questions it aims to answer are:

Does this procedure successfully reduce chronic heel pain as measured by the Visual Analog Scale (VAS) over 12 months?

How safe is the procedure, specifically regarding the frequency of serious medical problems or adverse events related to the device?

Participants will:

Undergo a minimally invasive procedure where a doctor uses a small tube (catheter) to inject a temporary blocking agent (LipioJoint) into specific blood vessels in the foot.

Receive a phone call one day after the procedure to check for early side effects.

Participate in four follow-up telehealth visits over the course of one year (at 1, 3, 6, and 12 months).

Complete pain intensity surveys (VAS) and report any changes in their use of other therapies or medications during these visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 25 years
* Subject provides written informed consent
* Patient with Plantar Fasciitis refractory to 3 months of conservative management
* Self reported pain of at least 4/10 on visual analog scale (VAS)
* Non-surgical candidate/looking to avoid surgery

Exclusion Criteria:

* Heel pain caused by acute fracture, recent trauma, inflammatory conditions, muscle/ligament injury, and etiologies related to bone mineral density.
* Steroid injection in the last 90 days from the embolization procedure
* Known severe allergy to Lipiodol and/or iodinated contrast media
* Diagnosis of peripheral arterial disease affecting the lower extremities
* Pregnancy or breastfeeding
* Anticoagulation or irreversible coagulopathy
* GFR <45 or Serum creatinine > 2.0 mg/dl
* Type 1 Diabetes Mellitus

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain Change | Baseline to 12 months
  Pain - measured via VAS at baseline, 1-month, 3-month, 6-month, and 12-month follow-up
Safety (rate of adverse events) | Baseline to 12 month follow-up
  Safety - Percentage of subjects without serious adverse events related to the medical device

CONTACTS AND LOCATIONS:
Locations (1):
- Joint and Vascular Institute, Libertyville, Illinois, United States